CLINICAL TRIAL: NCT01081028
Title: Connect® MM- The Multiple Myeloma Disease Registry
Status: Terminated | Type: Observational
Why Stopped: Business objectives have changed
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: Connect ® MM; CC-5013-MM-036 (Other: Sponsor); CA078-1009 (Other: Sponsor)
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; MM; disease registry; Connect®
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cohort 1: Patients enrolled between Sep 2009 and Nov 2011: Newly diagnosed multiple myeloma patients enrolled between Sep 2009 and Nov 2011.
  Interventions: Other: First-line therapy
- Cohort 2: Patients enrolled between December 2012 and mid-2016: Newly diagnosed multiple myeloma patients enrolled between Dec 2012 and mid-2016
  Interventions: Other: First-line therapy
- Cohort 3: Patients enrolled from 2023: Relapsed/Refractory multiple myeloma patients receiving second-line therapy
  Interventions: Drug: Second-line Multiple Myeloma treatments

INTERVENTIONS:
Other: First-line therapy — As prescribed by treating physician
  Groups: Cohort 1: Patients enrolled between Sep 2009 and Nov 2011; Cohort 2: Patients enrolled between December 2012 and mid-2016
Drug: Second-line Multiple Myeloma treatments — As prescribed by the treating physician
  Groups: Cohort 3: Patients enrolled from 2023

SUMMARY:
The purpose of the Connect® MM Registry is to explore the natural history and real world management of patients with newly diagnosed symptomatic multiple myeloma (MM) and provide unique insights into the management of MM and the impact of this hematologic disorder on patients.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 and 2

* Newly diagnosed with symptomatic MM within 2 months of enrollment in Connect® MM registry
* Age ≥18 years
* Willing and able to provide signed informed consent
* Agrees to complete patient assessment questionnaires either alone or with minimal assistance from caregivers and/or trained site personnel

Cohort 3

* Received 1L therapy for symptomatic active MM and subsequently has evidence of disease progression. Prior 1L MM treatment received, including anti-myeloma therapy, transplant, chemotherapy, radiation, and surgery, must be known.
* Initiated or intends to initiate 2L systemic therapy for MM after the first documented relapsed/refractory date (i.e. 1L PD).
* Enrollment date must be within 90 days of start date (or intended start date) of 2L systemic therapy.

Exclusion Criteria:

Cohort 1 and 2

- None

Cohort 3

* Patient's 1L MM treatment was for smoldering MM or MGUS, and not for symptomatic MM
* Currently active in any MM Registry, including but not limited to, the Connect® MM registry or another Celgene/BMS-Sponsored registry.
* Patients who have discontinued from Connect® MM or another Celgene/BMS-Sponsored registry could be considered for enrollment in Cohort 3, if inclusion and exclusion criteria are met.
* Currently enrolled or intending to enroll within 90 days in any interventional clinical trial in which any treatment is an investigational product that cannot be identified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed multiple myeloma and being treated in community or academic settings in the United States
Sampling Method: Non-Probability Sample
Enrollment: 3008 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Participant baseline demographics | Baseline
Participant medical history | Baseline
Participant Multiple Myeloma diagnosis information | Baseline
Participant Multiple Myeloma treatment history | Baseline
Multiple Myeloma-related supportive concomitant medications and procedures | Baseline, every 3-months up to 5 years (Cohort 3), or up to 16 years (Cohort 1 & 2), or date of early discontinuation
Occurance of second primary malignancy | Baseline, every 3-months up to 5 years (Cohort 3), or up to 16 years (Cohort 1 & 2), or date of early discontinuation
Number of participants enrolled in a clinical trial | Baseline, every 3-months up to 16 years or date of early discontinuation
  Cohort 1 and 2 only
Lines of therapy prescribed | Baseline, every 3-months up to 5 years (Cohort 3), or up to 16 years (Cohort 1 & 2), or date of early discontinuation
Participant disease response assessment results | Baseline, every 3-months up to 5 years (Cohort 3), or up to 16 years (Cohort 1 & 2), or date of early discontinuation

SECONDARY OUTCOMES:
Participant socioeconomic status | Baseline
  Cohort 3 only
Participant EuroQol-5 Dimensions (EQ-5D) questionnaire results | Baseline, every 3-months up to 5 years (Cohort 3) or up to 16 years (Cohort 1 and 2), or date of early discontinuation
Participant Functional Assessment of Cancer Therapy - Multiple Myeloma (FACT-MM) questionnaire results | Baseline, every 3-months up to 5 years (Cohort 3) or up to 16 years (Cohort 1 and 2), or date of early discontinuation
Participant Visual Analogue Score (VAS) questionnaire results | Baseline, every 3-months up to 5 years (Cohort 3) or up to 16 years (Cohort 1 and 2), or date of early discontinuation
Participant participant survival status | Every 3-months up to 5 years (Cohort 3) or up to 16 years (Cohort 1 and 2), or date of early discontinuation
Participant participant Adverse Events (AEs) | Every 3-months up to 5 years (Cohort 3) or up to 16 years (Cohort 1 and 2) or date of early discontinuation
Reason for registry discontinuation | Date of early discontinuation assessed up to 5 years (Cohort 3) or up to 16 years (Cohort 1 and 2)
Reason for treatment initiation or discontinuation | Baseline, and every 3-months up to 5 years or date of early discontinuation
  Cohort 3 only
Participant COVID-19 infection and vaccination status | Baseline, and every 3-months up to 5 years or date of early discontinuation
  Cohort 3 only
Treating clinician response to frailty questionnaire | Baseline, and every 3-months up to 5 years or date of early discontinuation
  Cohort 3 only
Participant Brief Pain Inventory (BPI) questionnaire results | Baseline, and every 3-months up to 5 years or date of early discontinuation
  Cohort 3 only
Participant response to social support questionnaire | Baseline, and every 3-months up to 5 years or date of early discontinuation
  Cohort 3 only
Treating clinician response to social support questionnaire | Baseline, and every 3-months up to 5 years or date of early discontinuation
  Cohort 3 only
Number of participants that have received stem cell transplant | Baseline, and every 3-months up to 5 years or date of early discontinuation
  Cohort 3 only
Number of hospitalization or emergency room visits | Every 3-months up to 5 years (Cohort 3) or up to 16 years (Cohort 1 and 2) or date of early discontinuation
Cause of death | Every 3-months up to 5 years (Cohort 3) or up to 16 years (Cohort 1 and 2) or date of early discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (253):
- United States (252):
  - The Cancer Center of Huntsville, Huntsville, Alabama
  - DCH Health System, Tuscaloosa, Alabama
  - US Oncology - Arizona Oncology Associates - Rudasill, Tucson, Arizona
  - St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Clopton Clinic Hematology/Oncology, Jonesboro, Arkansas
  - Little Rock Hematology Oncology Associates, PA, Little Rock, Arkansas
  - Pacific Cancer Medical Center, Inc, Anaheim, California
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Southbay Oncology Hematology Partners, Campbell, California
  - Compassionate Cancer Care Medical Group (Corona), Corona, California
  - Southwest Cancer Care, Escondido, California
  - Compassionate Cancer Care Medical Group (Fountain Valley), Fountain Valley, California
  - Virginia K. Crosson Cancer Center, Fullerton, California
  - TORI - Antelope Valley Cancer Center, Lancaster, California
  - Monterey Bay Oncology, Monterey, California
  - TORI - North Valley Hematology/Oncology, Northridge, California
  - Hematology Oncology Associates, Oakland, California
  - Comprehensive Cancer Center, Palm Springs, California
  - Bay Area Cancer Research Group, LLC, Pleasant Hill, California
  - New Hope Cancer & Research Institute, Pomona, California
  - Campassionate Cancer Care Medical Group (Riverside), Riverside, California
  - Capitol Hematology Oncology Medical Group - Sutter Roseville, Roseville, California
  - TORI - Central Coast Medical Oncology, Santa Maria, California
  - Redwood Regional Medical Group, Inc., Santa Rosa, California
  - Stockton Hematology Oncology Medical Group, Inc., Stockton, California
  - Institute for Myeloma and Bone Cancer Research, West Hollywood, California
  - US Oncology- Rocky Mountain Cancer Center-Aurora, Aurora, Colorado
  - US Oncology - Rocky Mountain Cancer Center-Boulder, Boulder, Colorado
  - US Oncology- Rocky Mountain Cancer Center at the Pavillion, Colorado Springs, Colorado
  - US Oncology - Rocky Mountain Cancer Center-Colorado Springs, Colorado Springs, Colorado
  - US Oncology - Rocky Mountain Cancer Center-Midtown, Denver, Colorado
  - US Oncology - Rocky Mountain Cancer Center-Rose, Denver, Colorado
  - TORI - St. Mary's Advanced Medical Pavilion, Grand Junction, Colorado
  - US Oncology - Rocky Mountain Cancer Center-Lakewood, Lakewood, Colorado
  - US Oncology - Rocky Mountain Cancer Center-Littleton, Littleton, Colorado
  - US Oncology - Rocky Mountain Cancer Center-Sky Ridge, Lone Tree, Colorado
  - US Oncology - Rocky Mountain Cancer Center-Longmont, Longmont, Colorado
  - US Oncology - Rocky Mountain Cancer Center-Parker, Parker, Colorado
  - US Oncology - Rocky Mountain Cancer Center-Thornton, Thornton, Colorado
  - Medical Specialists of Fairfield, Fairfield, Connecticut
  - Medical Oncology and Blood Disorders, LLP, Manchester, Connecticut
  - Hospital of Central Connecticut, New Britain, Connecticut
  - Hematology Oncology, PC, Stamford, Connecticut
  - Delaware Clinical & Laboratory Physicians, PA, Newark, Delaware
  - Hematology Oncology Associates, Boynton Beach, Florida
  - University Cancer Institute, Boynton Beach, Florida
  - Collaborative Research Group, Boynton Beach, Florida
  - Flora Research Associates, Coral Springs, Florida
  - Archbold Cancer Center, Deerfield Beach, Florida
  - Flora Research Associates, Deerfield Beach, Florida
  - Broward Oncology Associates, PA, Fort Lauderdale, Florida
  - Florida Cancer Specialists & Research Institute, Gainesville, Florida
  - Memorial Cancer Institute, Hollywood, Florida
  - US Oncology - Florida Cancer Institute - New Hope-Hudson, Hudson, Florida
  - Integrated Community Oncology Network, LLC, Jacksonville, Florida
  - Watson Clinic, Lakeland, Florida
  - Cancer & Blood Disease Center, Lecanto, Florida
  - Pasco Hernando Oncology Associates (Kumar), New Port Richey, Florida
  - US Oncology - Florida Cancer Institute - New Hope-New Port Richey, New Port Richey, Florida
  - Sacred Heart Medical Oncology Group, Pensacola, Florida
  - Cancer Care Centers of Brevard, Rockledge, Florida
  - Florida Hospital Waterman-Lake County Oncology & Hematology, The Villages, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Peachtree Hematology-Oncology Consultants, Atlanta, Georgia
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Summit Cancer Care, Savannah, Georgia
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Cancer Care & Hematology Specialists of Chicagoland, PC, Arlington Heights, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Univeristy of Chicago Medical Center, Section of Hematology/Oncology, Chicago, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Northshore University Health System, Evanston, Illinois
  - Ingalls Cancer Research Center, Harvey, Illinois
  - Joliet Oncology, Joliet, Illinois
  - Medical Arts Associates, Ltd, Moline, Illinois
  - Oncology Specialists, S.C., Niles, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Orchard Research, Skokie, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Indiana Blood and Marrow Transplant, LLC, Beech Grove, Indiana
  - St. Francis Cancer Research, Beech Grove, Indiana
  - Center for Cancer Care @ Goshen Health Systems, Goshen, Indiana
  - Indiana University Cancer Center Clinical Research Office, Indianapolis, Indiana
  - Cancer Research-Munster, Munster, Indiana
  - Cancer Care Center Inc., New Albany, Indiana
  - Oncology Hematology Associates of SW IN, Newburgh, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - McFarland Clinic, Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Iowa Blood and Cancer Care of PCI, Cedar Rapids, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Cedar Valley Medical Specialists, Waterloo, Iowa
  - Covenant Clinic, Waterloo, Iowa
  - Cancer Center of Kansas, PA, Wichita, Kansas
  - Baptist Hospital East, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Alliance Hematology Oncology, PA, Westminster, Maryland
  - Capecod Hospital/Davenport Mugar Cancer Center, Hyannis, Massachusetts
  - Fallon Clinic, Worcester, Massachusetts
  - Michigan State University/Bay Regional Medical Center, Bay City, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Michigan State University/McLaren Regional Medical Center, Flint, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Michigan State University/Breslin Cancer Center, Lansing, Michigan
  - Michigan State University/Lapeer Regional Medical Center, Lapeer, Michigan
  - Michigan State University/Mount Clemens Regional Medical Center, Mount Clemens, Michigan
  - Newland Medical Associates, Novi, Michigan
  - Michigan State University/Memorial Cancer Center, Owosso, Michigan
  - Newland Medical Associates, Southfield, Michigan
  - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Park Nicollet Institute - Louisiana Ave., Saint Louis Park, Minnesota
  - Jackson Oncology Associates, Jackson, Mississippi
  - St. Louis Cancer Care, LLP, Chesterfield, Missouri
  - Capitol Comprehensive Cancer Care Clinic, Jefferson City, Missouri
  - St. Joseph Oncology, Saint Joseph, Missouri
  - St. John's Medical Research Institute, Springfield, Missouri
  - University Hematology Oncology, Inc., St Louis, Missouri
  - Washington University in St. Louis, Division of Oncology, Section of Bone Marrow Transplantation & Leukemia, St Louis, Missouri
  - Hematology Oncology Consultants, Inc, St Louis, Missouri
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Montana Cancer Institute Foundation, Missoula, Montana
  - Nebraska Hematology Oncology, PC, Lincoln, Nebraska
  - Southeast Nebraska Hematology & Oncology Consultants, PC, Lincoln, Nebraska
  - TORI - Comprehensive Cancer Centers of NV, Henderson, Nevada
  - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - VA Sierra Nevada Healthcare System, Reno, Nevada
  - Essex Oncology of North Jersey, PA, Belleville, New Jersey
  - The Center for Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - Drs. Forte, Schleider, Attas & Condemi, PA, Englewood, New Jersey
  - Hematology-Oncology Associates of Northern NJ dba Carol G. Simon, Morristown, New Jersey
  - Steeplechase Cancer Center, Somerville, New Jersey
  - US Oncology - New York Oncology Hematology, PC-Albany, Albany, New York
  - US Oncology - Albany Medical Cancer Center, Albany, New York
  - US Oncology - Amsterdam Community Cancer Program, Amsterdam, New York
  - Jonah Cancer Care Center & ECMC, Buffalo, New York
  - US Oncology - Cavell Cancer Treatment Program, Hudson, New York
  - Broome Oncology, Johnson City, New York
  - Arena Oncology Associates, PC, Lake Success, New York
  - US Oncology - New York Oncology Hematology, PC-Latham, Latham, New York
  - US Oncology - New York Oncology Hematology, PC-Rexford, Rexford, New York
  - SUNY Upstate Medical University - Adult Program, Syracuse, New York
  - Bronx River Medical Associates, The Bronx, New York
  - Eastchester Center for Cancer Care, The Bronx, New York
  - US Oncology - Troy Cancer Treatment Program, Troy, New York
  - US Oncology - Cancer Centers of North Carolina - Cary, Cary, North Carolina
  - DUMC Division of Cellular Therapy/ABMT, Durham, North Carolina
  - Carolina Oncology Specialists, PA, Hickory, North Carolina
  - Emerywood Hematology/Oncology, High Point, North Carolina
  - US Oncology - Cancer Centers of North Carolina - Falls, Raleigh, North Carolina
  - Legacy Pharma Research, Bismarck, North Dakota
  - Med Center One, Bismarck, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Cancer Research Office, Akron, Ohio
  - Gabrail Cancer Center Research, Canton, Ohio
  - Cleveland VA Medical Center, Cleveland, Ohio
  - Mid Ohio Oncology/Hematology, Inc, Columbus, Ohio
  - Hematology Oncology Center, Inc, Elyria, Ohio
  - Lawrence M. Stallings MD LTD dba Trilogy Cancer Care, Wooster, Ohio
  - US Oncology - Willamette Valley Cancer Institute - Eugene, Eugene, Oregon
  - US Oncology - Willamette Valley Cancer Institute - Springfield, Springfield, Oregon
  - Oncology Hematology of Lehigh Valley, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Consultants in Medical Oncology and Hematology, PC, Drexel Hill, Pennsylvania
  - Andrews and Patel Associates, Harrisburg, Pennsylvania
  - US Oncology - Medical Oncology Associates (Nahar), Kingston, Pennsylvania
  - Lancaster Cancer Center, Lancaster, Pennsylvania
  - The Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - UPCI Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Berks Hematology Oncology Associates, Reading, Pennsylvania
  - Hematology & Oncology Associates of Rhode Island, Cranston, Rhode Island
  - Charleston Hematology Oncology Associates, PA, Charleston, South Carolina
  - US Oncology - Cancer Centers of the Carolinas - Easley, Easley, South Carolina
  - US Oncology - Cancer Centers of the Carolinas - Butternut, Greenville, South Carolina
  - US Oncology - Cancer Centers of the Carolinas - West Faris, Greenville, South Carolina
  - US Oncology - Cancer Centers of the Carolinas - Eastside, Greenville, South Carolina
  - SC Cancer Specialists, PA, Hilton Head Island, South Carolina
  - US Oncology - Cancer Center of the Carolinas - Seneca, Seneca, South Carolina
  - US Oncology - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Sanford Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Family Cancer Center, PLLC, Collierville, Tennessee
  - SCRI, Nashville, Tennessee
  - US Oncology - Texas Cancer Center - Abilene (South), Abilene, Texas
  - US Oncology - Texas Oncology, PA - Amarillo, Amarillo, Texas
  - US Oncology - Texas Oncology - Arlington South, Arlington, Texas
  - US Oncology - Texas Oncology - Midtown, Austin, Texas
  - US Oncology - Texas Oncology Cancer Center, Austin, Texas
  - US Oncology - South Austin Cancer Center, Austin, Texas
  - US Oncology - Texas Oncology North Austin, Austin, Texas
  - Austin Cancer Centers, Austin, Texas
  - US Oncology - Southwest Regional Cancer Center - North, Austin, Texas
  - US Oncology - Texas Oncology, PA - Bedford, Bedford, Texas
  - St. Joseph Regional Cancer Center, Bryan, Texas
  - US Oncology - Texas Oncology Cedar Park, Cedar Park, Texas
  - Scott & White Clinic, College Station, Texas
  - South Texas Institute of Cancer, Corpus Christi, Texas
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - US Oncology - Texas Cancer Center at Medical City, Dallas, Texas
  - US Oncology -Texas Oncology, PA - Dallas, Dallas, Texas
  - US Oncology - El Paso Cancer Treatment Ctr, El Paso, Texas
  - US Oncology - Texas Oncology, PA - Forth Worth, Fort Worth, Texas
  - US Oncology - Southwest Forth Worth Cancer Center, Fort Worth, Texas
  - US Oncology - Texas Oncology, PA - Garland, Garland, Texas
  - US Oncology - Texas Oncology - Grapevine, Grapevine, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - The Methodist Hospital Research Institute-AOCT, Houston, Texas
  - Southlake Oncology dba Las Colinas Hematology Oncology, Irving, Texas
  - US Oncology - San Antonio Tumor & Blood Clinic - Kerrville, Kerrville, Texas
  - US Oncology - Texas Oncology - Kyle, Kyle, Texas
  - US Oncology - Longview Cancer Center, Longview, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - US Oncology - Allison Cancer Center, Midland, Texas
  - US Oncology - Texas Oncology - Odessa, Odessa, Texas
  - US Oncology - North Texas Regional Cancer Center, Plano, Texas
  - US Oncology - Texas Oncology Plano West Cancer Center, Plano, Texas
  - US Oncology - Texas Oncology Seton Williamson, Round Rock, Texas
  - US Oncology - Texas Oncology - Round Rock Cancer Center, Round Rock, Texas
  - US Oncology - Cancer Care Centers of South Texas, San Antonio, Texas
  - US Oncology - HOAST - Medical Dr., San Antonio, Texas
  - US Oncology - San Antonio Tumor & Blood Clinic - M. Oak, San Antonio, Texas
  - US Oncology - Texas Oncology - San Marcos, San Marcos, Texas
  - Scott & White Healthcare Department of Research, Temple, Texas
  - ETMC dba Blood and Cancer Center - East Texas, Tyler, Texas
  - ETMC dba Tyler Hematology Oncology, Tyler, Texas
  - US Oncology - Texas Oncology Cancer Care and Research Center, Waco, Texas
  - US Oncology - Texoma Cancer Center, Wichita Falls, Texas
  - Central Utah Clinic, American Fork, Utah
  - Northern Utah Associates, Ogden, Utah
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah
  - US Oncology - Arlington Fairfax Hematology Oncology, Arlington, Virginia
  - US Oncology - Fairfax-Northern VA Hem-Onc PC, Fairfax, Virginia
  - US Oncology - Fairfax Northern Virginia Hematology-Oncology, PC-Gainesville, Gainesville, Virginia
  - US Oncology - Fairfax-Northern Virgina Hem-Onc, PC-Leesburg, Leesburg, Virginia
  - US Oncology - Shenandoah Oncology - Winchester, Winchester, Virginia
  - US Oncology - Fairfax-Northern Virginia Hem-Onc, PC-Woodbridge, Woodbridge, Virginia
  - Peace Health Medical Group, Bellingham, Washington
  - US Oncology - Puget Sound Cancer Center-Edmonds, Edmonds, Washington
  - Providence Everett Medical Center, Everett, Washington
  - Columbia Basin Hematology and Oncology, Kennewick, Washington
  - US Oncology - Puget Sound Cancer Center-Seattle, Seattle, Washington
  - US Oncology - Cancer Care Northwest - Sherman, Spokane, Washington
  - Medical Oncology Associates PS, Spokane, Washington
  - Providence St. Mary Regional Cancer Center, Walla Walla, Washington
  - US Oncology - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington
  - West Virginia University - Clinical Trials Research Unit, Morgantown, West Virginia
  - Fox Valley Hematology & Oncology, Appleton, Wisconsin
  - St. Vincent Hospital/Green Bay Oncology, Green Bay, Wisconsin
  - CMS Water Tower Medical Commons Medical Oncology #100, Milwaukee, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Auxilio Cancer Center, San Juan, Puerto Rico

REFERENCES:
- [Background] Rifkin RM, Jagannath S, Durie BGM, Narang M, Terebelo HR, Gasparetto CJ, Toomey K, Hardin JW, Wagner L, Parikh K, Abouzaid S, Srinivasan S, Kitali A, Zafar F, Abonour R. Treatment Outcomes and Health Care Resource Utilization in Patients With Newly Diagnosed Multiple Myeloma Receiving Lenalidomide-only Maintenance, Any Maintenance, or No Maintenance: Results from the Connect MM Registry. Clin Ther. 2018 Jul;40(7):1193-1202.e1. doi: 10.1016/j.clinthera.2018.05.017. Epub 2018 Jul 23. PMID 30007443
- [Background] Shah JJ, Abonour R, Gasparetto C, Hardin JW, Toomey K, Narang M, Srinivasan S, Kitali A, Zafar F, Flick ED, Rifkin RM. Analysis of Common Eligibility Criteria of Randomized Controlled Trials in Newly Diagnosed Multiple Myeloma Patients and Extrapolating Outcomes. Clin Lymphoma Myeloma Leuk. 2017 Sep;17(9):575-583.e2. doi: 10.1016/j.clml.2017.06.013. Epub 2017 Jun 17. PMID 28886839
- [Background] Terebelo HR, Abonour R, Gasparetto CJ, Toomey K, Durie BGM, Hardin JW, Jagannath S, Wagner L, Narang M, Flick ED, Srinivasan S, Yue L, Kitali A, Agarwal A, Rifkin RM; CONNECT MM Registry Investigators. Development of a prognostic model for overall survival in multiple myeloma using the Connect(R) MM Patient Registry. Br J Haematol. 2019 Dec;187(5):602-614. doi: 10.1111/bjh.16139. Epub 2019 Aug 5. PMID 31382320
- [Result] Rifkin RM, Abonour R, Terebelo H, Shah JJ, Gasparetto C, Hardin J, Srinivasan S, Ricafort R, Nagarwala Y, Durie BG. Connect MM Registry: The Importance of Establishing Baseline Disease Characteristics. Clin Lymphoma Myeloma Leuk. 2015 Jun;15(6):368-76. doi: 10.1016/j.clml.2014.12.002. Epub 2014 Dec 11. PMID 25617035
- [Result] Rifkin RM, Abonour R, Shah JJ, Mehta J, Narang M, Terebelo H, Gasparetto C, Toomey K, Hardin JW, Lu JJ, Kenvin L, Srinivasan S, Knight R, Nagarwala Y, Durie BG. Connect MM(R) - the Multiple Myeloma Disease Registry: incidence of second primary malignancies in patients treated with lenalidomide. Leuk Lymphoma. 2016 Sep;57(9):2228-31. doi: 10.3109/10428194.2015.1132419. Epub 2016 Jan 13. No abstract available. PMID 26766599
- [Result] Terebelo H, Srinivasan S, Narang M, Abonour R, Gasparetto C, Toomey K, Hardin JW, Larkins G, Kitali A, Rifkin RM, Shah JJ. Recognition of early mortality in multiple myeloma by a prediction matrix. Am J Hematol. 2017 Sep;92(9):915-923. doi: 10.1002/ajh.24796. Epub 2017 Jul 19. PMID 28543165
- [Result] Jagannath S, Abonour R, Durie BGM, Gasparetto C, Hardin JW, Narang M, Terebelo HR, Toomey K, Wagner L, Srinivasan S, Kitali A, Yue L, Flick ED, Agarwal A, Rifkin RM. Heterogeneity of Second-Line Treatment for Patients With Multiple Myeloma in the Connect MM Registry (2010-2016). Clin Lymphoma Myeloma Leuk. 2018 Jul;18(7):480-485.e3. doi: 10.1016/j.clml.2018.04.007. Epub 2018 May 4. PMID 29844008
- [Result] Jagannath S, Abonour R, Durie BGM, Narang M, Terebelo HR, Gasparetto CJ, Toomey K, Hardin JW, Wagner L, Agarwal A, Srinivasan S, Kitali A, Flick ED, Sturniolo M, Rifkin RM. Impact of post-ASCT maintenance therapy on outcomes in patients with newly diagnosed multiple myeloma in Connect MM. Blood Adv. 2018 Jul 10;2(13):1608-1615. doi: 10.1182/bloodadvances.2018017186. PMID 29986853
- [Result] Abonour R, Wagner L, Durie BGM, Jagannath S, Narang M, Terebelo HR, Gasparetto CJ, Toomey K, Hardin JW, Kitali A, Gibson CJ, Srinivasan S, Swern AS, Rifkin RM. Impact of post-transplantation maintenance therapy on health-related quality of life in patients with multiple myeloma: data from the Connect(R) MM Registry. Ann Hematol. 2018 Dec;97(12):2425-2436. doi: 10.1007/s00277-018-3446-y. Epub 2018 Jul 29. PMID 30056582
- [Result] Jagannath S, Rifkin RM, Gasparetto CJ, Toomey K, Durie BGM, Hardin JW, Terebelo HR, Wagner L, Narang M, Ailawadhi S, Omel JL, Srinivasan S, He M, Ung B, Kitali A, Flick ED, Agarwal A, Abonour R; CONNECT MM Registry Investigators. Treatment Journeys of Patients With Newly Diagnosed Multiple Myeloma (NDMM): Results From The Connect MM Registry. Clin Lymphoma Myeloma Leuk. 2020 May;20(5):272-276. doi: 10.1016/j.clml.2019.10.002. Epub 2019 Oct 14. No abstract available. PMID 32144027
- [Result] Ailawadhi S, Jagannath S, Lee HC, Narang M, Rifkin RM, Terebelo HR, Durie BGM, Toomey K, Hardin JW, Gasparetto CJ, Wagner L, Omel JL, He M, Yue L, Flick ED, Agarwal A, Abonour R; Connect MM Registry Investigators. Association between race and treatment patterns and survival outcomes in multiple myeloma: A Connect MM Registry analysis. Cancer. 2020 Oct 1;126(19):4332-4340. doi: 10.1002/cncr.33089. Epub 2020 Jul 24. PMID 32706404
- [Result] Abonour R, Rifkin RM, Gasparetto C, Toomey K, Durie BGM, Hardin JW, Terebelo HR, Jagannath S, Narang M, Ailawadhi S, Omel JL, Lee HC, Srinivasan S, Kitali A, Agarwal A, Wagner L; CONNECT MM Registry Investigators. Effect of initial treatment on health-related quality of life in patients with newly diagnosed multiple myeloma without immediate stem cell transplant intent: results from the Connect(R) MM Registry. Br J Haematol. 2021 Apr;193(1):93-100. doi: 10.1111/bjh.17131. Epub 2020 Oct 29. PMID 33118614
- [Derived] Ailawadhi S, Lee HC, Omel J, Toomey K, Hardin JW, Gasparetto CJ, Jagannath S, Rifkin RM, Durie BGM, Narang M, Terebelo HR, Joshi P, Jou YM, Mouro J, Yu E, Abonour R. Impact of lenalidomide-bortezomib-dexamethasone induction on patients with newly diagnosed multiple myeloma and renal impairment: Results from the Connect(R) MM Registry. Blood Cancer J. 2024 Nov 11;14(1):198. doi: 10.1038/s41408-024-01177-6. PMID 39528478
- [Derived] Lee HC, Ramasamy K, Weisel K, Abonour R, Hardin JW, Rifkin RM, Ailawadhi S, Terebelo HR, Durie BGM, Tang D, Joshi P, Liu L, Jou YM, Che M, Hernandez G, Narang M, Toomey K, Gasparetto C, Wagner LI, Jagannath S. Treatment Patterns, Survival, Quality of Life, and Healthcare Resource Use Among Patients With Triple-Class Refractory Multiple Myeloma in US Clinical Practice: Findings From the Connect MM Disease Registry. Clin Lymphoma Myeloma Leuk. 2023 Feb;23(2):112-122. doi: 10.1016/j.clml.2022.11.008. Epub 2022 Nov 23. PMID 36567211
- [Derived] Engelhardt M, Ihorst G, Singh M, Rieth A, Saba G, Pellan M, Lebioda A. Real-World Evaluation of Health-Related Quality of Life in Patients With Multiple Myeloma From Germany. Clin Lymphoma Myeloma Leuk. 2021 Feb;21(2):e160-e175. doi: 10.1016/j.clml.2020.10.002. Epub 2020 Oct 24. PMID 33218965
- [Derived] Ailawadhi S, Jagannath S, Narang M, Rifkin RM, Terebelo HR, Toomey K, Durie BGM, Hardin JW, Gasparetto CJ, Wagner L, Omel JL, Kumar V, Yue L, Kitali A, Agarwal A, Abonour R; Connect MM Registry Investigators. Connect MM Registry as a national reference for United States multiple myeloma patients. Cancer Med. 2020 Jan;9(1):35-42. doi: 10.1002/cam4.2656. Epub 2019 Nov 7. PMID 31701679